CLINICAL TRIAL: NCT05242887
Title: Validation of the 3-Minute Diagnostic Interview for CAM-defined Delirium (3D-CAM) and the Ultra-Brief CAM (UB-CAM) in French.
Brief Title: Validation of the 3D-CAM and the UB-CAM in French
Acronym: French-UB-CAM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0903; 2021-A02130-41 (Other: IDRCB)
Record Dates: First submitted 2022-02-07; First posted 2022-02-16 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Delirium
Keywords: Delirium; CAM; UB-CAM; 3D-CAM
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults hospitalized in acute geriatric units: Response to a questionnaire
  Interventions: Diagnostic Test: Delirium screening using 3D-CAM and UB-CAM

INTERVENTIONS:
Diagnostic Test: Delirium screening using 3D-CAM and UB-CAM — Patients will be evaluated with 3D-CAM and UB-CAM by a trained examiner (geriatrician, resident or neuropsychologist). On the same day, they will be given a reference diagnosis of delirium based on DSM-V criteria by another trained examiner, blind to the results of the UB-CAM and 3D-CAM.

SUMMARY:
Delirium is very common in hospitalized older patients and associated with serious clinical bad outcomes (e.g. increased risk of functional decline and death). Despite its high prevalence in the hospital setting, delirium remains underdiagnosed. A better identification would allow an early management and a reduction of its complications.

The validation of easy-to-use and quick and formalized tools for the identification of delirium and their implementation in the clinical practice are necessary.

Recently, the 3D-CAM (3-minutes Diagnostic interview for Confusion Assessment Method -defined delirium) and the UB-CAM (Ultra-Brief CAM) showed very high sensitivity and specificity (> 90%), compared to the reference standard (Diagnostic and Statistical Manual of Mental Disorders (DSM criteria)) for the diagnosis of delirium.

The investigators aimed to evaluate the sensitivity and specificity of the French versions of the 3D-CAM and the UB-CAM used in delirium screening in older adults hospitalized in geriatric units, compared to reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Adults hospitalized in acute geriatric units
* Aged 65 or older
* Patient (or relative) not objecting to participating in the study

Exclusion Criteria:

- Legal protection regimes (guardianship, curatorship)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults hospitalized in acute geriatric units
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of the performance of a rapid diagnostic tool (UB-CAM) for acute confusional state, translated into French | At inclusion
  Presence or absence of a confusional state (with UB-CAM and the gold standard: DSM-V criteria)

SECONDARY OUTCOMES:
Evaluation of the time taken to use this tool | At inclusion
  Completion time (minutes, seconds)
Evaluation of the diagnostic performance of another diagnostic tool (3D-CAM), already translated into French | At inclusion
  Presence or absence of a confusional state (with 3D-CAM and the gold standard: DSM-V criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine GARNIER-CRUSSARD, MD, MSc, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital des Charpennes, Institut du Vieillissement, Hospices Civils de Lyon, Villeurbanne, Lyon, France

IPD SHARING:
Plan to Share IPD: No